CLINICAL TRIAL: NCT04373213
Title: Evaluation of the Fluid Response of SARS-CoV-2 (COVID-19) Patients in Intensive Care; Pleth Variability Index
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Erzincan University (Other)
Responsible Party: Principal Investigator, ILKE KUPELI, assoc. prof., Erzincan University
Other Study IDs: EBYU COVİD PVI
Record Dates: First submitted 2020-04-30; First posted 2020-05-04 (Actual); Last update posted 2020-05-04 (Actual); Status verified 2020-04

CONDITIONS: Pleth Variability Index

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Pleth variability index: Patients undergoing fluid management with Pleth variability index
  Interventions: Diagnostic Test: Pleth variability index
- hemodynamic: Patients undergoing fluid management with hemodynamic findings
  Interventions: Diagnostic Test: Pleth variability index

INTERVENTIONS:
Diagnostic Test: Pleth variability index — The usefulness of Pleth variability index in predicting fluid response in patients with COVID 19

SUMMARY:
In this study; We aimed to investigate the role of pleth variability index, which is a noninvasive method, in showing fluid response in SARS-CoV-2 (COVID-19) patients, which we know is appropriate fluid management.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized in COVID 19 anesthesia intensive care unit
* Patients over the age of 18

Exclusion Criteria:

* Patients under the age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years of age who have been hospitalized in the COVID 19 anesthesia intensive care unit
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-05-05 (Estimated); Primary Completion 2020-06-05 (Estimated); Study Completion 2020-06-15 (Estimated)

PRIMARY OUTCOMES:
Pleth variability index | 1 month
  Pleth variability index levels

CONTACTS AND LOCATIONS:
Overall Officials: ILKE KUPELI, Principal Investigator — Dr.
Locations (1):
- Erzincan University, Erzincan, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Basso F, Berdin G, Virzi GM, Mason G, Piccinni P, Day S, Cruz DN, Wjewodzka M, Giuliani A, Brendolan A, Ronco C. Fluid management in the intensive care unit: bioelectrical impedance vector analysis as a tool to assess hydration status and optimal fluid balance in critically ill patients. Blood Purif. 2013;36(3-4):192-9. doi: 10.1159/000356366. Epub 2013 Dec 20. PMID 24496190
- [Background] Claure-Del Granado R, Mehta RL. Fluid overload in the ICU: evaluation and management. BMC Nephrol. 2016 Aug 2;17(1):109. doi: 10.1186/s12882-016-0323-6. PMID 27484681
- [Result] de Oliveira OH, Freitas FG, Ladeira RT, Fischer CH, Bafi AT, Azevedo LC, Machado FR. Comparison between respiratory changes in the inferior vena cava diameter and pulse pressure variation to predict fluid responsiveness in postoperative patients. J Crit Care. 2016 Aug;34:46-9. doi: 10.1016/j.jcrc.2016.03.017. Epub 2016 Mar 30. PMID 27288609
- [Result] Piskin O, Oz II. Accuracy of pleth variability index compared with inferior vena cava diameter to predict fluid responsiveness in mechanically ventilated patients. Medicine (Baltimore). 2017 Nov;96(47):e8889. doi: 10.1097/MD.0000000000008889. PMID 29382017
- [Result] Liu T, Xu C, Wang M, Niu Z, Qi D. Reliability of pleth variability index in predicting preload responsiveness of mechanically ventilated patients under various conditions: a systematic review and meta-analysis. BMC Anesthesiol. 2019 May 8;19(1):67. doi: 10.1186/s12871-019-0744-4. PMID 31068139